CLINICAL TRIAL: NCT05795569
Title: Removal of Nasogastric Feeding Tube Post Extubation in ICU : a Prospective Randomized Trial
Acronym: FIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRO-2022-15; 2022-A02605-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Deglutition Disorders; Intensive Care Unit Syndrome; Swallowing Disorder; Feeding or Eating Disorder
MeSH Terms: conditions — Deglutition Disorders; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Intervention Group: Nasogastric tube removal upon extubation with protocolized PED screening Control Group: Conventional nasogastric tube management and PED screening strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Procedure: Nasogastric Tube removal during extubation; Diagnostic Test: Yale Swallow Protocol
- Control Group (Active Comparator)
  Interventions: Procedure: Classif Nasogastric Tube Management; Diagnostic Test: Classic swallowing test

INTERVENTIONS:
Procedure: Nasogastric Tube removal during extubation — The nurse in charge of the patient and under the cover of a medical prescription, will proceed to the systematic removal of the nasogastric tube during the extubation procedure
  Arms: Intervention Group
Diagnostic Test: Yale Swallow Protocol — The dysphagia will be evaluated in a systematic way between 1 hour and 6 hours post-extubation with the help of the "Yale Swallow Protocol" (YSP) by the caregivers trained to the passing of the "YSP" (nurse or physiotherapist or ICU doctor).
  Arms: Intervention Group
Procedure: Classif Nasogastric Tube Management — The removal of the nasogastric tube will not be performed during the extubation procedure and the time of removal will be left to the discretion of the attending physician (as currently performed in the unit).
  Arms: Control Group
Diagnostic Test: Classic swallowing test — Post-extubation dysphagia will be assessed as we do in the unit. Currently, the caregivers in charge of the patient do a gel water test "Nutrisens Hydra'Fruit level 4" when the attending physician prescribes it.
  Arms: Control Group

SUMMARY:
Post-extubation dysphagia (PED) is a frequent but still underestimated condition in the intensive care units (ICU). In the international literature, the manifestations and consequences of PED lead to intra- and post-intensive care comorbidities.

The exact etiology of PED is unknown, but considered multifactorial. Numerous causes, acquired during ICU, can lead to a delay in the reintroduction of intravenous nutrition, or even favor the development of inhalation pneumopathy. One of these causes is the presence of the nasogastric tube.

The incidence of ECD varies from 3 to 62%. Its presence impacts morbidity and mortality. Preventive strategies for PED have only been studied with questionable methodologies.

The goal of ICU therapists is to detect PED as early as possible in order to implement curative strategies such as adapted nutrition and early swallowing rehabilitation.

DETAILED DESCRIPTION:
There are several tools available to diagnose PED. These assessment methods are numerous and not subject to consensus.

There are expensive instrumental methods requiring experts, which allow for accurate diagnosis but cannot be routinely used at the ICU patient's bed. For the ICU patient, bed-side clinical assessments seem more appropriate.

The "Yale swallow protocol" (YSP), is the most used test in the literature. Its sensitivity in predicting PED at 96.5%, a negative predictive value of 97.9% and a false negative rate of less than 2%, seem to make it the most suitable.

Currently, no recommendations have been made by French or international ICU societies on the appropriate time or method for PED assessment.

Regarding the treatment of PED, the literature shows that physiotherapy management would not significantly reduce its incidence, nor accelerate the resumption of per os feeding.

No study has examined the impact of nasogastric tube removal combined with the use of a standardized swallow test on post-extubation ECD.

For all these reasons, we plan to evaluate the interventional strategy consisting in removing the nasogastric feeding tube as soon as extubation, to carry out between 1 hour and 6 hours post extubation the "Yale swallow protocol", to allow a resumption of feeding as soon as possible while screening the dysphagic patients.

The research hypothesis is therefore:

"Systematic removal of the nasogastric tube during the extubation procedure associated with an early swallow test in the ICU allows an early per-os nutritional resumption in comparison with the classical strategy of nasogastric tube management and swallowing disorders assessment"

ELIGIBILITY:
Inclusion Criteria:

* Extubation prescribed by the attending physisian
* Intubation for more than 48 hours
* Presence of a nasogastric tube
* RASS score equal to 0 at the time of screening.

Exclusion Criteria:

* Gastric tube for gastric emptying (suction or bag)
* Inability to remain alert for prolonged periods of time for the swallow test
* Pre-existing dysphagia
* Patient fed by nasogastric tube or jejunostomy before ICU stay
* Tracheostomized patient
* Contraindication to a bed head elevation > 30°.
* Contraindication to the resumption of feeding
* Pregnant or breastfeeding woman
* Decision to limit active therapies
* Protected person (under guardianship or curatorship) / Person under court protection
* Person not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Time to feeding resumption post extubation | Day 1
  If the patient passes the YSP or the classic swallowing test, a per-os diet resumption will be started and we will record the time of passing the test as the time of per-os feeding resumption.

SECONDARY OUTCOMES:
Reintubation rate | Day 7
  Defined as the necessity to intubate a patient when he/she was once extubated during his/her stay.
Rate of acquired pneumonia in the intensive care unit | Day 28
  Defined as a new pneumonia acquired after the first extubation
Weight loss during ICU stay | Day 28
  Defined as the difference between admission and discharge weight
Undernutrition status | Day 7
  Defined as the blood pre-albumin level
ICU lenght of stay | Day 28
  Defined as the number of days of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Cecile FOSSAT, Pt, Principal Investigator — CHR Orleans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntyre M, Doeltgen S, Dalton N, Koppa M, Chimunda T. Post-extubation dysphagia incidence in critically ill patients: A systematic review and meta-analysis. Aust Crit Care. 2021 Jan;34(1):67-75. doi: 10.1016/j.aucc.2020.05.008. Epub 2020 Jul 29. PMID 32739246
- [Background] Leder SB, Warner HL, Suiter DM, Young NO, Bhattacharya B, Siner JM, Davis KA, Maerz LL, Rosenbaum SH, Marshall PS, Pisani MA, Siegel MD, Brennan JJ, Schuster KM. Evaluation of Swallow Function Post-Extubation: Is It Necessary to Wait 24 Hours? Ann Otol Rhinol Laryngol. 2019 Jul;128(7):619-624. doi: 10.1177/0003489419836115. Epub 2019 Mar 6. PMID 30841709
- [Background] Zuercher P, Moser M, Waskowski J, Pfortmueller CA, Schefold JC. Dysphagia Post-Extubation Affects Long-Term Mortality in Mixed Adult ICU Patients-Data From a Large Prospective Observational Study With Systematic Dysphagia Screening. Crit Care Explor. 2022 Jun 8;4(6):e0714. doi: 10.1097/CCE.0000000000000714. eCollection 2022 Jun. PMID 35765374
- [Background] Warner HL, Suiter DM, Nystrom KV, Poskus K, Leder SB. Comparing accuracy of the Yale swallow protocol when administered by registered nurses and speech-language pathologists. J Clin Nurs. 2014 Jul;23(13-14):1908-15. doi: 10.1111/jocn.12340. Epub 2013 Sep 6. PMID 24033866